CLINICAL TRIAL: NCT05984628
Title: Umbilical Cord Stem Cells for Skin Grafts in Donor Site Wounds
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, ChenXiaosong, Director of Plastic Surgery and Regenerative Medicine, Fujian Medical University Union Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020GXB001-01
Record Dates: First submitted 2023-07-14; First posted 2023-08-09 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Skin Wound; Scar, Hypertrophic
Keywords: hUCMSC; Skin Wound; Scar, Hypertrophic; Stem cell
MeSH Terms: conditions — Cicatrix, Hypertrophic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The efficacy evaluation component is conducted in a blinded manner, meaning that the assessors of efficacy outcomes are composed of plastic surgeons who are not members of the research team, have not participated in the intervention, and are unaware of the group allocation of the patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- human umbilical cord mesenchymal stem cells (Experimental): Injection of human umbilical cord mesenchymal stem cells (hUCMSC) into the donor site.
  1. Dosage of stem cell preparation: Calculated based on the area of the donor site, with a cell count of 1X10^5cells/cm2.
  2. Administration method: The cells are prepared as an injectable suspension using a blank solvent for stem cells at a concentration of 1X10^6 cells/ml (0.1 ml/cm2).
  3. Timing of administration: Administered immediately after completion of the donor site harvesting procedure.
  4. Treatment duration: The stem cell administration is a single dose, administered at the specified timing as described above
  Interventions: Procedure: human umbilical cord mesenchymal stem cells
- blank solvent (Placebo Comparator): Injection of an equal volume of blank solvent for suspension of stem cells into the donor site.
  1. Dosage of Control group preparation: Calculated based on the area of the donor site.
  2. Administration method: Injection of an equal volume of blank solvent for suspension of stem cells into the donor site.
  3. Timing of administration: Administered immediately after completion of the donor site harvesting procedure.
  4. Treatment duration: The Control group administration is a single dose, administered at the specified timing as described above
  Interventions: Procedure: blank solvent

INTERVENTIONS:
Procedure: human umbilical cord mesenchymal stem cells — After the completion of the donor site harvesting in the experimental group, allogeneic umbilical cord mesenchymal stem cells are injected into the deep layer of the de-epithelialized area and the surrounding 0.5cm subcutaneous region. After the injection, the wound is covered and dressed with conventional dressings.
  Arms: human umbilical cord mesenchymal stem cells
Procedure: blank solvent — After the completion of the donor site harvesting in the experimental group, the de-epithelialized area and the surrounding 0.5cm subcutaneous region is injected an equal volume of blank solvent for stem cell suspension in the control group. After the injection, the wound is covered and dressed with conventional dressings.
  Arms: blank solvent

SUMMARY:
The goal of this clinical trial is to evaluate the safety and effectiveness of human umbilical cord mesenchymal stem cell (hUCMSC) therapy in patients undergoing medium-thickness skin grafts for donor site wounds. The study aims to answer the following main questions:

* Question 1: Does hUCMSC therapy improve the healing quality and speed of donor site wounds in comparison to standard treatment?
* Question 2: Does hUCMSC therapy reduce scar formation in the donor site wounds?

Participants in this study will undergo medium-thickness skin grafts, and those in the treatment group will receive hUCMSC therapy. The main tasks for participants will involve regular follow-up visits, monitoring of wound healing progress, and assessment of any potential side effects or complications associated with the therapy.

In order to evaluate the effectiveness of hUCMSC therapy, researchers will compare the treatment group receiving hUCMSC therapy with a control group that receives standard treatment alone. The aim is to determine if the use of hUCMSC therapy leads to improved healing outcomes and reduced scar formation compared to the standard treatment group.

DETAILED DESCRIPTION:
The donor site of the medium-thickness skin graft procedure usually forms scars or even hypertrophic scars, which significantly differ from normal skin physiology and cause discomfort to patients such as itching and burning sensations. Currently, the pathological mechanism of scar formation is not fully understood. There is a pressing clinical need for new methods to improve the healing quality and speed of donor site wounds in patients undergoing medium-thickness skin grafts and to reduce scar formation.

It is well known that various types of stem cells from different sources are involved in the process of wound repair. Under the regulation of various signaling molecules and chemotactic factors, they migrate to the wound, proliferate, and differentiate into various cellular components of the skin, thus constructing new tissue structures and achieving wound healing. Stem cells possess powerful self-renewal and multi-directional differentiation abilities. Some stem cells have been successfully applied in the treatment of severe burn wounds and non-healing wounds, yielding promising results.

Furthermore, in recent years, tissue engineering techniques have been used to combine stem cells with appropriate scaffolds to create tissue-engineered skin, utilizing the potential of stem cells for multi-directional differentiation and rapid expansion. This approach allows for rapid coverage and functional reconstruction of large-area wounds. Therefore, we also hope to enhance the healing quality of donor site wounds in patients undergoing medium-thickness skin grafts and inhibit excessive scar formation by utilizing stem cell technology.

Among the various options, the use of human umbilical cord mesenchymal stem cells (UCMSC) is highly feasible for treating donor site wounds in medium-thickness skin graft procedures. UCMSC has abundant sources, easy collection, easy expansion, no harm to donors, no ethical controversies, potential for industrialization and standardized clinical treatment, and excellent biological characteristics.

This study aims to investigate the safety and efficacy of human umbilical cord mesenchymal stem cell (hUCMSC) therapy for donor site wounds in medium-thickness skin grafts, as well as its effect in reducing scar formation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18 and 60 years old with extensive scars, large benign tumors, or fresh wounds on the body surface.
2. Patients who undergo medium-thickness skin graft surgery (donor site can be from the thigh, abdomen, or back).
3. Participants who have a thorough understanding of the study objectives, significance, implementation plan, potential benefits, risks involved, measures to address risks, and the rights and obligations of the subjects (including privacy protection and the right to withdraw), and are willing to participate in this clinical study and can cooperate effectively.

Exclusion Criteria:

Participants who meet any of the following criteria are not suitable for inclusion:

1. Hypertension, hypotension, heart disease (including history of myocardial ischemia, coronary heart disease, myocarditis).
2. Liver or kidney dysfunction.
3. Infectious diseases (including viral hepatitis, syphilis, HIV/AIDS, etc.).
4. Venous thrombosis, thoracic or abdominal aortic aneurysm, aortic dissection.
5. Blood disorders (abnormal coagulation function, anemia, leukemia, polycythemia vera, aplastic anemia, etc.).
6. Allergic conditions (urticaria, bronchial asthma, history of allergic reactions to two or more drugs or foods).
7. Respiratory system diseases (chronic bronchitis, emphysema, bronchiectasis, respiratory failure, chronic obstructive pulmonary disease, interstitial pneumonia).
8. Digestive system diseases (severe gastric or duodenal ulcers, chronic gastritis, chronic pancreatitis).
9. Urinary system diseases (chronic urinary tract infections, nephritis, nephrotic syndrome).
10. Endocrine system diseases (hyperthyroidism, diabetes, acromegaly, pituitary diseases, adrenal diseases, diabetes insipidus).
11. Organic neurological disorders or psychiatric illnesses (encephalitis, sequelae of traumatic brain injury, epilepsy, schizophrenia, hysteria, depression, severe insomnia, neurasthenia).
12. Chronic skin diseases (especially infectious, allergic, and inflammatory systemic skin diseases, such as extensive eczema, pemphigus, pemphigoid).
13. Autoimmune diseases and collagen diseases (such as systemic lupus erythematosus, dermatomyositis, scleroderma).
14. History of long-term smoking, alcohol abuse, or drug addiction.
15. History of major surgeries (such as gastric, lung, splenic, renal, or liver resection).
16. History of other significant malignant tumors.
17. Blood donation or organ transplantation within the past 5 years.
18. Pregnancy, lactation, menstrual period, or within 1 year after termination of pregnancy.
19. Previous circumstances of being rejected for voluntary blood donation.
20. Other situations deemed unsuitable for participation in this study by the investigators.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
Time to epithelialization of the skin wound | 12 months
  Record the size of the donor site wound at each follow-up time point and document it with photographs.
Observation of scar formation | 12 months
  Record the height and erythema of the donor site scar at each follow-up time point and document them with photographs.
  It will be assessed using, Vancouver scar scale at time of presentation and at 12 months after the intervention. Pre and post intervention ratings will be compared and percentage increase or decrease in the rating will be documented. Vancouver Scar Scale is a 13 points scale and includes four parameters, pigmentation, vascularity pliability and height of scar.13 It is an objective scale and examining doctor will assess and record score out of 13. Lesser the score better is the scar

SECONDARY OUTCOMES:
Itching at wound site | 12 months
  It will be assessed at the time of presentation and at 12 months after the intervention using severity of pruritus scale. It is 4 point rating scale from 0 (no itch) to 3(severe itch disturbing the sleep) assessing severity of pruritus within 24-hours recall period. Pre and post intervention ratings will be compared and percentage increase or decrease in the rating will be documented.
Pain At scar Site | 12 months
  Patient will be asked to rate his/her current, best and worst pain level over past 24 hours on scale of 0 (no pain) to 10 (worst pain imaginable). Pain at scar site will be assessed at time of presentation and then at 12 months after start of the treatment. Pre and post intervention ratings will be compared and percentage increase or decrease in the rating will be documented. This scale is chosen due to its high feasibility and good compliance.

CONTACTS AND LOCATIONS:
Overall Officials: xiaosong xiaosong, xiaosong, Study Chair — Affiliated Union Hospital of Fujian Medical University
Locations (1):
- Chenxiaosong, Fujian, Fuzhou, China